CLINICAL TRIAL: NCT03580538
Title: The Short-term Effects of a Resistive Training Program Using Elastic Tubing in Cardiac Patients: Clinical Trial
Brief Title: Training With Elastic Tubing in Cardiopaths: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mayara Moura Alves da Cruz, physiotherapist, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44443915.5.0000.5515
Record Dates: First submitted 2018-06-14; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Resistance Training; Muscular Strength; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elastic tube group (Experimental)
  Interventions: Other: resistive exercise with elastic tube

INTERVENTIONS:
Other: resistive exercise with elastic tube — performed training with elastic tubing for six weeks, twice a week and the load was progressively increased every 15 days.

SUMMARY:
Background: Resistance training is effective in cardiac rehabilitation; however, other types of training, such as elastic tubing, are rarely used and may present good therapeutic alternatives. Due to its practicality and cost effectiveness, training using elastic tubing may become an important tool in cardiovascular rehabilitation. Objective: To evaluate muscular strength, functional capacity, aerobic capacity and quality of life in patients with cardiovascular diseases in phase II of rehabilitation, after resistance training with elastic tubing. Methods: patients with cardiovascular diseases performed training with elastic tubing for six weeks, twice a week and the load was progressively increased every 15 days. The following muscle groups were evaluated and trained: shoulder abductors and flexors, elbow flexors, and knee flexors and extensors. Muscular strength was evaluated using a dynamometer; functional capacity with a 6-minute walk test and ergospirometric test; and quality of life using the SF-36 questionnaire. Data normality was assessed using the Shapiro Wilk test. Comparisons before and after training were performed using the paired Student's t test or the Wilcoxon test (p <5%).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Aged between 45-79 years
* Clinical diagnosis of heart disease (coronary artery disease, postoperative myocardial revascularization, acute myocardial infarction)
* In phase II of CRP for at least three months

Exclusion Criteria:

* Patients hemodynamically unstable
* Patients with changes in medication for a minimum of 30 days
* Patients who presented arteriopathies, neurological, muscular or orthopedic disorders, such as rheumatism and unstable heart disease that could be detected by electrocardiogram, and lung diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Muscular Strength at 6 weeks | The evaluation of muscular strength was performed at the start of the intervention protocol and after 6 weeks.
  The evaluation of muscular strength was performed at the start of the intervention protocol and after 6 weeks, using a digital force gauge, brand Force Gauge®, model FG-100kg - United States, and all results were expressed in Newtons (N). The evaluation was performed with the dominant member of each patient, using a steel cord coated with rigid plastic attached to a dynamometer, with one end attached to a fixed bar and the other end to the distal portion of the dominant member of the patient
Change from baseline Functional Capacity at 6 weeks | was performed at the start of the intervention protocol and after 6 weeks
  The evaluation of functional capacity was carried out through the 6-minute walk test (6MWT). The 6MWT followed the criteria established by the American Thoracic Society15. The test was performed in a gym hall at Oeste Paulista University, Presidente Prudente/SP-Brazil, and was repeated twice with an interval of 30 minutes between attempts and the highest value was taken into account, during the test Standardized verbal performance incentives were given every minute. During the 6MWT was measured blood pressure, oximetry, perception subjective of effort, heart and respiratory rate.
Change from baseline Evaluation of maximal aerobic capacity at 6 weeks | was performed at the start of the intervention protocol and after 6 weeks
  The patients underwent a cardiopulmonary test performed by a cardiologist. All tests were performed on a treadmill (Inbrasport ATL 2000). The modified Bruce protocol16 was used and the test performed until voluntary exhaustion. No patient presented alterations in the electrocardiogram that prevented the realization and completion of the test.
  Cardiovascular parameters were monitored continuously: heart rate through the Polar S810i, Finland, arterial oxygen saturation using the Mindray PM 50 pulse oximeter, Brazil, and the subjective perception of effort.17 The ventilatory variables were obtained through the VO2000 gas analyzer (Medical Graphics, USA) calibrated before each test according to the manufacturer's instructions. The average air flow was used in all tests and obtained every 10 seconds, Aerograph®, Michigan, USA.
Change from baseline Evaluation of quality of life at 6 weeks | was performed at the start of the intervention protocol and after 6 weeks
  The quality of life of these patients was assessed using the generic quality of life evaluation questionnaire SF-36, validated in Brazil, which has eight dimensions that are scored from 0 to 100. For each dimension, values greater than 50 are positive in relation to a good perception of quality of life

IPD SHARING:
Plan to Share IPD: Undecided